CLINICAL TRIAL: NCT06290895
Title: The Effect of Artificial Oocyte Activation on Blastocysts Rate in Patients With Low Fertilization Rate
Brief Title: Artificial Oocyte Activation
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3465
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Infertility; Ovarian Insufficiency
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- In-vitro fertilization (IVF) cycle using artificial oocyte activation (AOA)
  Interventions: Other: women having had a second IVF cycle with AOA
- In-vitro fertilization (IVF) cycle without artificial oocyte activation (AOA)

INTERVENTIONS:
Other: women having had a second IVF cycle with AOA — The absence of synergy between the oocyte and sperm leads to a negative impact on oocyte activation. Physiological oocyte activation requires a sperm-derived enzyme called phospholipase C zeta to cause the release of calcium in the form of oscillations from internal storages.
  Groups: In-vitro fertilization (IVF) cycle using artificial oocyte activation (AOA)

SUMMARY:
Studies reported that calcium signal deficiency or insufficiency during oocyte activation are related with embryo arrest and blastocyst quality. The utilization of Artificial Oocyte Activation (AOA) is safe and does not increase birth defects, cognition, language and motor skills. AOA is the first line of treatment in patients with globozoospermia (round headed spermatozoa). Poor responders in in-vitro fertilization (IVF) cycles represent a major challenge for fertility specialists and comprises about 10-15% of patients undergoing controlled ovarian hyperstimulation. The absence of synergy between the oocyte and sperm leads to a negative impact on oocyte activation. The European Society of Human and REproduction (ESHRE) recommends AOA in cases with failed fertilization/ low fertilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with poor or no blastocyst development in their primary cycle
* Group 1 - second cycle using AOA following the poor blastocyst development cycle
* Group 2 - second cycle without AOA following the poor development cycle

Exclusion Criteria:

* All cycles who do not have repeat cycles following the poor blastocyst development cycle

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women able to have oocyte retrieval after in-vitro fertilization
Study Population: Data spreadsheet from 2018 to 2023 of patients having undergone an IVF cycle
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Blastocyst rate | 5 days after oocyte fertilization
  Likelihood of an oocyte fertilized to blastocyst stage

CONTACTS AND LOCATIONS:
Overall Officials: Simon Phillips, PhD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No